CLINICAL TRIAL: NCT05283928
Title: Implant Primary Stability and Ridge Dimensional Changes Utilizing the Osseodensification Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Popi Stylianou, Clinical Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-21-0597
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Dental Implants
Keywords: osseodensification; ridge expansion
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: Each participant served as their own control. Each participant had at least 1 control implant and at least 1 test implant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- OsseoDensification (OD) protocol (Experimental)
  Interventions: Device: OsseoDensification (OD) protocol
- standard drilling (SD) protocol (Active Comparator)
  Interventions: Device: standard drilling (SD) protocol (NobelReplace® Conical)

INTERVENTIONS:
Device: OsseoDensification (OD) protocol — Osseodensification is a drilling process by which bone is being compacted and auto-grafted in an outwardly expanding direction from the osteotomy. When the osseodensification drills are being rotated in a reversed, non-cutting direction a strong and dense layer of bone is formed along the walls and base of the osteotomy.
  Arms: OsseoDensification (OD) protocol
Device: standard drilling (SD) protocol (NobelReplace® Conical) — osteotomy preparation through bone excavation is necessary in implant site development for the placement of dental implants. The process involves a forward cutting process with removal of bone tissue creating appropriate size osteotomy for the dental implant.
  Arms: standard drilling (SD) protocol

SUMMARY:
The purpose of this study is to compare ridge dimensional changes between densification and standard drilling protocols and to compare primary and secondary stability of implants placed by bone densification and standard drilling protocols

ELIGIBILITY:
Inclusion Criteria:

* Patients who understand and agree to this study.
* Adequate Oral hygiene
* One or more edentulous spaces, which are 10 weeks or longer after extractions

Exclusion Criteria:

* Pregnancy.
* Smoking of more than 5 cigarettes/day.
* History of alcoholism or drug abuse during the last 5 years.
* Uncontrolled Hypertension or diabetes.
* Patient with malignant tumor.
* Patients on daily dose of steroids.
* Patients with history of chemotherapy or radiation for the last 12 months.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Popi Stylianou, DDS,MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 participants were enrolled. Each participant served as their own control. Each participant had at least 1 control implant and at least 1 test implant
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Started | 15; 20 Implants | 15; 20 Implants
Completed | 15; 20 Implants | 15; 20 Implants
Not Completed | 0; 0 Implants | 0; 0 Implants

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: The purpose of this study is to compare ridge dimensional changes between densification and standard drilling protocols and to compare primary and secondary stability of implants placed by bone densification and standard drilling protocols.
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.67 (14.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Ridge Width at Crest
Description: bone ridge width will be measured using a Caliper
Time Frame: day of implant surgery
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Implants
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 15 | 15
Number analyzed (Implants) | 20 | 20
millimeters | 0.84 (0.59) | 0.01 (0.45)

2. Primary Outcome: Change in Bone Ridge Width at 5mm Apical From Crest
Description: bone ridge width will be measured using a Caliper
Time Frame: day of implant surgery
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Implants
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 15 | 15
Number analyzed (Implants) | 20 | 20
millimeters | 0.62 (0.65) | 0.11 (0.64)

3. Primary Outcome: Change in Bone Ridge Width at 10mm Apical From Crest
Description: bone ridge width will be measured using a Caliper
Time Frame: day of implant surgery
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Implants
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 15 | 15
Number analyzed (Implants) | 20 | 20
millimeters | 0.29 (0.76) | 0.01 (0.46)

4. Secondary Outcome: Primary Stability of the Implants as Measured by the Insertion Torque Values
Description: Insertion torque refers to the force used to insert an implant into bone, and it is reported in units of Newton-Centimeters (N-cms).
Time Frame: day of implant surgery
Measure: Mean (Standard Deviation); unit: Newton-centimeters
Units Other Than Participants: Implants
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 15 | 15
Number analyzed (Implants) | 20 | 20
Newton-centimeters | 57.7 (23.4) | 45 (25.5)

5. Secondary Outcome: Primary Stability of the Implants as Indicated by the Implant Stability Quotient (ISQ) as Measured by the Resonance Frequency Analysis Using the Ostell ISQ Meter Baseline(After Implant Placement)
Description: The Implant Stability Quotient (ISQ) value is a measurement used to assess the stability of dental implants. It is obtained by resonance frequency analysis and ranges from 1 to 100, with higher values indicating greater stability.
Time Frame: baseline(after implant placement)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 15 | 15
Number analyzed (Implants) | 20 | 20
score on a scale | 73.7 (7.23) | 67.0 (8.26)

6. Secondary Outcome: Primary Stability of the Implants as Indicated by the Implant Stability Quotient (ISQ) as Measured by the Resonance Frequency Analysis Using the Ostell ISQ Meter 3 Weeks After Implant Placement
Description: as for outcome 5
Time Frame: 3 weeks after implant placement
Population: Noting that some participants had multiple implants, data for 6 implants in the OsseoDensification (OD) protocol arm were not collected, which includes data for 4 participants. Noting that some participants had multiple implants, data for 6 implants in the standard drilling (SD) protocol arm were not collected, which includes data for 4 participants
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 11 | 11
Number analyzed (Implants) | 14 | 14
score on a scale | 75 (6.87) | 69.8 (7.99)

7. Secondary Outcome: Primary Stability of the Implants as Indicated by the Implant Stability Quotient (ISQ) as Measured by the Resonance Frequency Analysis Using the Ostell ISQ Meter 6 Weeks After Implant Placement
Description: as for outcome 5
Time Frame: 6 weeks after implant placement
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 11 | 11
Number analyzed (Implants) | 14 | 14
score on a scale | 75.3 (6.16) | 70.8 (9.25)

8. Secondary Outcome: Primary Stability of the Implants as Indicated by the Implant Stability Quotient (ISQ) as Measured by the Resonance Frequency Analysis Using the Ostell ISQ Meter 12 Weeks After Implant Placement
Description: as for outcome 5
Time Frame: 12 weeks after implant placement
Population: Data for 1 implant in the OsseoDensification (OD) protocol arm were not collected, including 1 participant for whom no implant data were collected. Data for 1 implant in the standard drilling (SD) protocol arm were not collected, including 1 participant for whom no implant data were collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 14 | 14
Number analyzed (Implants) | 19 | 19
score on a scale | 76.8 (5.18) | 73.3 (7.31)

9. Secondary Outcome: Volume of the Ridge as Assessed by the Cone Beam Computer Tomography (CBCT)
Time Frame: 6 months post implantation
Population: Data were not collected for this outcome measure.
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percent Change of Buccal Bone Thickness as Assessed by the Cone Beam Computer Tomography at 1.5 mm From the Implant Platform
Description: The buccal bone thickness (BBT) was measured using cone beam computed tomography (CBCT). The percentage change in BBT was calculated by comparing the post-implant measurements to baseline values, with positive percentages indicating an increase in thickness and negative percentages indicating a decrease in thickness.
Time Frame: 6 months post implantation
Population: Noting that some participants had multiple implants, data for 3 implants in the OsseoDensification (OD) protocol arm were not collected, which includes data for 2 participants. Noting that some participants had multiple implants, data for 3 implants in the standard drilling (SD) protocol arm were not collected, which includes data for 2 participants
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: Implants
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 13 | 13
Number analyzed (Implants) | 17 | 17
percent change | 6.24 (31.8) | -21.3 (20.3)

11. Secondary Outcome: Percent Change of Buccal Bone Thickness as Assessed by the Cone Beam Computer Tomography at 5 mm From the Implant Platform
Description: as for outcome 10
Time Frame: 6 months post implantation
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: Implants
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
Number analyzed (Participants) | 13 | 13
Number analyzed (Implants) | 17 | 17
percent change | 8.61 (25.3) | -15.1 (21.6)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | OsseoDensification (OD) Protocol | Standard Drilling (SD) Protocol
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT05283928/Prot_SAP_000.pdf